CLINICAL TRIAL: NCT00056511
Title: Comparing Effects of 3 Sources of Garlic on Serum Lipids
Brief Title: Comparing Effects of 3 Sources of Garlic on Cholesterol Levels
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: Office of Dietary Supplements (ODS) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01AT001108-01 (NIH)
Record Dates: First submitted 2003-03-14; First posted 2003-03-18 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Hypercholesterolemia
Keywords: Garlic; Supplements; Adults; Hypercholesterolemics; Randomized Clinical Trial
MeSH Terms: conditions — Hypercholesterolemia

INTERVENTIONS:
Drug: Fresh garlic or garlic supplements

SUMMARY:
The purpose of this study is to determine whether fresh garlic can positively affect cholesterol in adults with moderately high cholesterol levels. This study will also determine whether the same effects can be found for two main types of garlic supplements: a dried powdered garlic (designed to yield the same effect as fresh garlic) and an aged garlic extract preparation.

DETAILED DESCRIPTION:
Garlic supplements are the most consumed herbal products in the United States. The most common health claim made for garlic supplements is cholesterol lowering activity. This claim has not been supported by recent clinical trials and meta-analyses. However, data suggest that it is not necessarily the garlic that has been ineffective, but rather the particular garlic preparations being used. To date, the predominant type of garlic preparation used in these clinical trials has been dried garlic powders. A few clinical trials have reported beneficial lipid effects using an aged garlic extract, and only a small number of inconclusive uncontrolled trials have used fresh garlic. A rigorous trial directly comparing different types of garlic preparations for their effects on serum lipids is needed.

Adults with moderately elevated low density lipoprotein cholesterol (LDL-C) will be randomized to one of four groups for 6 months: fresh garlic, dried powdered garlic tablets, aged garlic extract tablets, or placebo control. The fresh garlic will be provided to patients with "study sandwiches"; all other groups will receive the same study sandwiches without the garlic. All patients will take daily study tablets, but the tablet assignment will be double-blind. Patients will pick up study sandwiches twice a week and study tablets once every 2 weeks for 28 weeks. Blood samples will be taken once a month, with additional blood draws at the start and end of the study.

ELIGIBILITY:
Inclusion Criteria:

* LDL-C 130-190 mg/dL (fasting single sample)
* BMI (body mass index) 19-30 kg/m2 (42-66 lb/m2)
* Weight stable for last 2 months
* Not actively on a weight loss plan
* Ethnicity representative of local population
* No plans to move from the area over the next 9 months

Exclusion Criteria:

* Pregnant, lactating, within 6 months postpartum, or planning to become pregnant in the next year
* Diabetes (type I or II) or history of gestational diabetes
* Heart disease
* Active neoplasms
* Renal or liver disease
* Hyperthyroidism or hypothyroidism
* Lipid lowering medications (known to affect lipid metabolism, platelet function, or antioxidant status)
* Blood pressure medications
* Excessive alcohol intake (self reported, more than 3 drinks/day)
* Currently under psychiatric care or severely clinically depressed

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220
Dates: Start 2002-05; Study Completion 2005-04

PRIMARY OUTCOMES:
LDL-cholesterol; measured at baseline, once a month, and post-intervention

SECONDARY OUTCOMES:
HDL-cholesterol; measured at baseline, once a month, and post-intervention
Triacylglycerols; measured at baseline, once a month, and post-intervention
Blood pressure; measured at baseline, once a month, and post-intervention
Platelet aggregation; measured at baseline, once a month, and post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D. Gardner, Ph.D., Principal Investigator — Stanford Center for Research in Disease Prevention
Locations (1):
- Stanford Center for Research in Disease Prevention, Palo Alto, California, United States

REFERENCES:
- [Derived] Gardner CD, Lawson LD, Block E, Chatterjee LM, Kiazand A, Balise RR, Kraemer HC. Effect of raw garlic vs commercial garlic supplements on plasma lipid concentrations in adults with moderate hypercholesterolemia: a randomized clinical trial. Arch Intern Med. 2007 Feb 26;167(4):346-53. doi: 10.1001/archinte.167.4.346. PMID 17325296